CLINICAL TRIAL: NCT01489462
Title: Strength Training for ARthritis Trial
Acronym: START
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01AR059105 (NIH); 1R01AR059105-01A1 (NIH)
Record Dates: First submitted 2011-11-22; First posted 2011-12-09 (Estimated); Last update posted 2020-04-20 (Actual); Status verified 2017-10

CONDITIONS: Knee Osteoarthritis
Keywords: Arthritis; Osteoarthritis; Strength Training
MeSH Terms: conditions — Osteoarthritis, Knee; Arthritis; Osteoarthritis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- High Intensity Strength Training (Experimental): The strength-training intervention will consist of 5-min warm-up, 40-min training, and 15-min cool-down. The 60-min sessions will be conducted 3 times/wk for 18 months. Every 2 weeks the load lifted will be adjusted so that the participants in this group are lifting 3 sets of each exercise at 75-90% of 1RM.
  Interventions: Behavioral: High Intensity Strength Training
- Low Intensity Strength Training (Experimental): The strength-training intervention will consist of 5-min warm-up, 40-min training, and 15-min cool-down. The 60-min sessions will be conducted 3 times/wk for 18 months. Every 2 weeks the load lifted will be adjusted so that the participants are lifting 3 sets of 15 repetitions at 30-40% of 1RM.
  Interventions: Behavioral: Low Intensity Strength Training
- Attention Control (Active Comparator): Participants in the control group will attend 60-min organized workshops 2 times/month for the first 6 months and then 1 time/month for months 7-18. Over the 18 months interactive presentations will cover such topics as foot care, nutrition, managing medication, and sleep practices, and experts will give wide-ranging lectures.
  Interventions: Behavioral: Attention Control

INTERVENTIONS:
Behavioral: High Intensity Strength Training — The strength-training intervention will consist of 5-min warm-up, 40-min training, and 15-min cool-down. The 60-min sessions will be conducted 3 times/wk for 18 months. Every 2 weeks the load lifted will be adjusted so that the participants in this group are lifting 3 sets of each exercise at 75-90% of 1RM.
  Arms: High Intensity Strength Training
Behavioral: Low Intensity Strength Training — The strength-training intervention will consist of 5-min warm-up, 40-min training, and 15-min cool-down. The 60-min sessions will be conducted 3 times/wk for 18 months. Every 2 weeks the load lifted will be adjusted so that the participants are lifting 3 sets of 15 repetitions at 30-40% of 1RM.
  Arms: Low Intensity Strength Training
Behavioral: Attention Control — Participants in the control group will attend 60-min organized workshops 2 times/month for the first 6 months and then 1 time/month for months 7-18. Over the 18 months interactive presentations will cover such topics as foot care, nutrition, managing medication, and sleep practices, and experts will give wide-ranging lectures.
  Arms: Attention Control

SUMMARY:
The primary purpose of this study is to compare the effects of a high and low intensity strength training programs vs. a control group on knee pain and compressive joint forces.

DETAILED DESCRIPTION:
Muscle loss and fat gain contribute to the disability, pain, and morbidity associated with knee osteoarthritis (OA), and thigh muscle weakness is an independent and modifiable risk factor for it. However, while all published treatment guidelines, supported by Level-1 evidence, recommend muscle strengthening to combat sarcopenia and improve muscle quality in knee OA patients, previous strength-training studies either used intensities or loads below recommended levels or were generally short, lasting only 6 to 24 weeks. Consequently, they had low-to-modest effect sizes, could not detect changes in disease progression, did not address underlying OA mechanisms, and provided little lasting clinical benefit. The positive effects of long-term, structured exercise are known to persist even years after supervised treatment terminates.

The efficacy of high intensity strength training in improving OA symptoms, slowing progression, and affecting the underlying mechanisms has not been examined due to the unsubstantiated belief that it might exacerbate symptoms. Our preliminary data clearly show excellent tolerance for high-intensity strength training as well as reduced pain and increased function among older adults with knee OA. Similar studies in healthy older adults found improvements in thigh muscle mass and decreases in thigh fat mass with minimal alteration in total body weight after 16-18 weeks of training. We now propose an 18-month, high-intensity strength-training intervention for older adults with knee OA, focused on improving thigh composition (more muscle and less fat). We hypothesize that in addition to short-term clinical benefits, combining greater duration with high intensity will alter thigh composition sufficiently to attain long-term changes in knee-joint forces, decrease inflammatory cytokines, lower pain levels, and slow OA progression, which has yet to be convincingly demonstrated for any OA treatment. These are important benefits that are not achievable with shorter interventions.

Participants will be randomized to one of 3 groups: high-intensity strength training; low-intensity strength training; or attention control. The primary clinical aim is to compare the interventions' effects on knee pain, and the primary mechanistic aim is to compare their effects on knee-joint compressive forces during walking, a mechanism that affects the OA disease pathway. Secondary aims will compare intervention effects on additional clinical measures of disease severity (e.g., function, mobility); disease progression, measured by xray; thigh muscle and fat volume, measured by CT; components of thigh muscle function, including hip abductor strength and quadriceps strength, power, and proprioception; additional measures of knee-joint loading; and inflammatory and OA biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Mild to Moderate Knee Osteoarthritis

Exclusion Criteria:

* BMI <20 kg/m2 and ≥45 kg/m2
* Knee varus malalignment
* Participation in formal strength training for more than 30 min/week in the past 6 months.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 377 (Actual)
Dates: Start 2012-03; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
WOMAC Pain | Baseline, 18 months
  To determine if an 18-month, high-intensity strength-training intervention significantly decreases pain relative to low-intensity strength training and attention control groups. The pain index assesses participants' pain on a scale, ranging from 0 (none) to 4 (extreme). The pain subscale consists of 5 items and total scores can range from 0-20, with larger scores indicating greater pain.
Knee Compressive Forces | Baseline, 18 Months
  To compare the effects of 18 months of high-intensity strength training, low-intensity strength training, and attention control on knee-joint compressive forces during walking.

SECONDARY OUTCOMES:
WOMAC Pain | Baseline, 6 months
  To determine if 6 months of high-intensity strength training reduces pain significantly more than 6 months of low-intensity strength training or an attention control. The pain index assesses participants' pain on a scale, ranging from 0 (none) to 4 (extreme). The pain subscale consists of 5 items and total scores can range from 0-20, with larger scores indicating greater pain.
WOMAC Function | Baseline, 6 months
  To determine if 6 months of high-intensity strength training improves function significantly more than 6 months of low-intensity strength training or an attention control. The LK version asks participants to indicate on a scale from 0 (none) to 4 (extreme) the degree of difficulty experienced in the last week due to knee OA. Individual scores for the 17 items are totaled to generate a summary score that could range from 0-68, with higher scores indicating poorer function.
Mobility | Baseline, 6 months
  To determine if 6 months of high-intensity strength training improves mobility significantly more than 6 months of low-intensity strength training or an attention control. Participants are told to walk as far as possible in 6 minutes on an established course.
Knee Compressive Forces | Baseline, 6 months
  To determine if 6 months of high-intensity strength training reduces knee-joint compressive loads significantly more than 6 months of low-intensity strength training or an attention control.
WOMAC Function | Baseline, 18 Months
  To compare the long-term effects of a high-intensity strength training, low-intensity strength training, and attention control group on function (clinical outcome). The LK version asks participants to indicate on a scale from 0 (none) to 4 (extreme) the degree of difficulty experienced in the last week due to knee OA. Individual scores for the 17 items are totaled to generate a summary score that could range from 0-68, with higher scores indicating poorer function.
Mobility | Baseline, 18 Months
  To compare the long-term effects of a high-intensity strength training, low-intensity strength training, and attention control group on mobility (clinical outcome). Participants are told to walk as far as possible in 6 minutes on an established course.
Knee Joint Loads | Baseline, 18 Months
  To compare the long-term effects of a high-intensity strength training, low-intensity strength training, and attention control group on knee joint loads (knee adductor moment, knee AP shear force) (mechanistic outcome).
Structural Outcomes | Baseline, 18 Months
  To compare the effects of 18-month, high-intensity strength training, low-intensity strength training, and attention control on OA progression by changes in x-ray (e.g., joint space width).
Thigh Composition & Muscle Function | Baseline, 18 Months
  To compare the effects on thigh muscle and fat volume of 18-month, high-intensity strength training, low-intensity strength training, and an attention control. To compare the effects of the interventions on components of muscle function, including hip abductor and quadriceps strength, and muscle power.
Inflammatory & OA Markers | Baseline, 6 Months, 18 Months
  To compare the effects of the interventions on inflammation markers (IL-6, TNFα, sTNFR1, leptin) and OA biomarkers (serum PIIANP, COMP, urinary levels of CTX-II).

CONTACTS AND LOCATIONS:
Overall Officials: Stephen P Messier, PhD, Principal Investigator — Wake Forest University
Locations (1):
- Wake Forest University, Winston-Salem, North Carolina, United States

REFERENCES:
- [Derived] Messier SP, Mihalko SL, Beavers DP, Nicklas BJ, DeVita P, Carr JJ, Hunter DJ, Lyles M, Guermazi A, Bennell KL, Loeser RF. Effect of High-Intensity Strength Training on Knee Pain and Knee Joint Compressive Forces Among Adults With Knee Osteoarthritis: The START Randomized Clinical Trial. JAMA. 2021 Feb 16;325(7):646-657. doi: 10.1001/jama.2021.0411. PMID 33591346
- [Derived] Messier SP, Mihalko SL, Beavers DP, Nicklas BJ, DeVita P, Carr JJ, Hunter DJ, Williamson JD, Bennell KL, Guermazi A, Lyles M, Loeser RF. Strength Training for Arthritis Trial (START): design and rationale. BMC Musculoskelet Disord. 2013 Jul 15;14:208. doi: 10.1186/1471-2474-14-208. PMID 23855596